CLINICAL TRIAL: NCT04029012
Title: A Pilot Study to Assess Efficacy and Safety of Methoxyflurane for Pain Control During Convective Thermal Therapy Using Rezūm System in Benign Prostatic Hyperplasia (BPH)
Brief Title: Penthrox in Rezūm BPH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dean Elterman (Other)
Responsible Party: Sponsor-Investigator, Dean Elterman, Clinician Investigator/ Urologist, Can-Am HIFU Inc.
Organization: Can-Am HIFU Inc. (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Penthrox in Rezūm BPH
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Pain; BPH
MeSH Terms: conditions — Pain | interventions — Methoxyflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Penthrox (Experimental): methoxyflurane inhaler (Penthrox) to be used 5 minutes (+/- 1 minutes) before procedure, and continuously breathing in the inhaler throughout the procedure.
  Interventions: Drug: Methoxyflurane

INTERVENTIONS:
Drug: Methoxyflurane — Methoxyflurane inhaler before Rezum procedure
  Other Names: Penthrox

SUMMARY:
Open-labeled, single-centre study

DETAILED DESCRIPTION:
Patients who have elected Convective Thermal Therapy using Rezūm System for the management of their BPH and fulfilled inclusion and exclusion criteria will sign informed consent form for the study. Patient will use Methoxyflurane inhaler (Penthrox™) on top of standard oral analgesia including oral lorazepam, oral Percocet® (oxycodone and acetaminophen) or oxycodone immediate-release, and intra-urethral lidocaine gel (Xylocaine®). Intravenous propofol will be used as rescue analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects of ≥ 18 years of age
* Patient who has elected Convective Thermal Therapy using Rezūm System for the management of their benign prostatic hyperplasia.
* No contra-indication on using Methoxyflurane inhaler (Penthrox™).
* Willing and able to accurately complete the required questionnaires.
* Willing and able to provide signed and dated informed consent.

Exclusion Criteria:

* Ongoing use of analgesic agents for chronic pain.
* Concomitant use of nephrotoxic agents.
* INR > 4.
* Use of Methoxyflurane inhaler (Penthrox™) within the previous 3 months.
* Known allergy to Lorazepam, Percocet/ Oxycodone, or Xylocaine® gel.
* Known personal or familial hypersensitivity to Methoxyflurane inhaler (Penthrox™) or other halogenated anesthetics.
* Clinically significant respiratory depression, cardiovascular instability, renal or hepatic impairment.
* An altered level of consciousness, due to any cause, including head injury, drugs, or alcohol.
* Known or genetically susceptible to malignant hyperthermia or a history of severe adverse reactions in either patient or relatives.
* A history of liver dysfunction after previous Methoxyflurane inhaler (Penthrox™) use or other halogenated anesthetics.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient with BPH
Enrollment: 10 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
Pain intensity | immediately after final injection of Rezūm treatment
  Visual Analog Scale (VAS) from the range of 0-10 (0 represents no pain, 10 represents maximum pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Can-Am HIFU Inc, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided